CLINICAL TRIAL: NCT07384988
Title: The Impact of Nitrous Oxide Sedation on Dental Fear and Anxiety Scores in Children Aged 6-10 Years: A Randomized Controlled Clinical Trial
Brief Title: The Impact of Nitrous Oxide Sedation on Dental Fear and Anxiety Scores in Children Aged 6-10 Years
Acronym: N₂O
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaoxing Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Xu Renjie, Sub-Investigator, Shaoxing Maternity and Child Health Care Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023SKY097
Record Dates: First submitted 2026-01-08; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Dental Anxiety
Keywords: Dental anxiety; Nitrous Oxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): The control group received only conventional local anesthesia and psychological comfort measures. Preoperatively, medical staff communicated thoroughly with the child and guardian to explain the treatment process and precautions, alleviating anxiety. The child's oral and systemic health was assessed to determine treatment difficulty. During treatment, articaine (Septodont, France) were administered under strict aseptic techniques to minimize pain. Continuous psychological support was provided through gentle communication, encouraging gestures, and distraction techniques such as soothing music or storytelling to help the child relax and cooperate. Postoperatively, the child was observed for any adverse reactions before being discharged with their guardian.
  Interventions: Behavioral: psychological support
- experimental group (Experimental): The experimental group received nitrous oxide anesthesia using a professional dental nitrous oxide inhalation sedation system (Matrx, the United States). This system featured precise gas concentration adjustment, real-time patient vital sign monitoring, and a reliable alarm system to ensure accurate, safe, and stable nitrous oxide administration.
  Interventions: Drug: Nitrous Oxide Sedation

INTERVENTIONS:
Drug: Nitrous Oxide Sedation — After the child was seated in the dental chair, an appropriately sized nasal mask was selected to ensure a secure fit without leakage. The child initially inhaled 100% oxygen for 3-5 minutes to adapt to the breathing pattern and eliminate nitrogen from the lungs. Nitrous oxide was then introduced at an initial concentration of 10%-15%, with adjustments made in increments of 5%-10% based on the child's anxiety level, treatment stimuli, and vital signs. Each adjustment was followed by 1-2 minutes of observation until the desired level of sedation was achieved.
  Arms: experimental group
Behavioral: psychological support — gentle communication, encouraging gestures, and distraction techniques such as soothing music or storytelling to help the child relax and cooperate.
  Arms: control group

SUMMARY:
Dental anxiety (DA) is highly prevalent among children undergoing dental procedures, with 50-80% experiencing fear that disrupts treatment and exacerbates oral health outcomes. While nitrous oxide (N₂O) sedation is widely used for its anxiolytic properties, evidence remains limited regarding its standardized efficacy in reducing pediatric fear and anxiety scores.

DETAILED DESCRIPTION:
This study adopted a randomized controlled trial (RCT) design, strictly adhering to the CONSORT (Consolidated Standards of Reporting Trials) guidelines to ensure scientific rigor, reliability, and transparency.The sample size was calculated based on previous literature and preliminary pilot study results. Referring to the standard deviations of dental fear and anxiety scores in similar studies, the significance level (α) was set at 0.05, and the power (1 - β) was set at 0.85 (90% power). With an effect size of 0.4, the study anticipated significant differences in fear and anxiety scores between the experimental and control groups. Using statistical formulas and considering practical constraints, the estimated sample size required for each group was no fewer than 58 participants to ensure sufficient statistical power.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged 6-10 years; 2.Classified as American Society of Anesthesiologists (ASA) physical status I-II; 3.Required dental treatments such as caries filling, pulp therapy, or tooth extraction; 4.Informed consent obtained from the child's guardian.

Exclusion Criteria:

* 1.Contraindications to nitrous oxide inhalation, such as severe cardiopulmonary dysfunction, intestinal obstruction, or pneumothorax; 2.Mental illness or intellectual disability that would hinder cooperation with assessments or treatment; 3.Received dental sedation or general anesthesia within the past month;

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
MDAS | From enrollment to the end of treatment at 1 week
  The Modified Dental Anxiety Scale, zero is equivalent to no anxiety and 5 indicates the worst possible anxiety, participants achieved a response if they scored a performance status of 0 on a scale ranging from 0 (best outcome) to 5 (worst outcome)
Behavioral Observation Scale | From enrollment to the end of treatment at 1 week
  The Frankl behavior rating scale was used to assess the children's behavior during treatment. This 4-point scale categorizes behavior , participants achieved a response if they scored a performance status of 1 on a scale ranging from 1 (best outcome) to 4 (worst outcome)
CFSS-DS | From enrollment to the end of treatment at 1 week
  Children's Fear Survey Schedule-Dental Subscale, participants achieved a response if they scored a performance status of 1 on a scale ranging from 1 (best outcome) to 5 (worst outcome)

SECONDARY OUTCOMES:
HR | immediately after the intervention
  heart rate
BP | systolic and diastolic will be assessed immediately after the intervention
  blood pressure
RR | immediately after the intervention
  respiratory rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoxing Maternity and Child Health Care Hospital, Shaoxing, Zhejiang, China